CLINICAL TRIAL: NCT03154593
Title: Prevalence and Impact of Chronic Oedema in a Population of Patients Prior to and Following Bariatric Surgery
Brief Title: Prevalence of Chronic Oedema in Obese Patients
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 16031
Record Dates: First submitted 2017-05-05; First posted 2017-05-16 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-07

CONDITIONS: Chronic Oedema; Obesity
Keywords: Prevalence
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: Stage 1 will determine the prevalence of chronic oedema among patients attending weight management services at the Royal Derby Hospital and how it impacts on every day life.
- Stage 2: Stage 2 will determine whether bariatric surgery improves the oedema.
  Interventions: Other: Stage 2 - Bariatric Surgery

INTERVENTIONS:
Other: Stage 2 - Bariatric Surgery — This observational study follows patients after routine bariatric surgery.
  Groups: Stage 2

SUMMARY:
Persistent swelling (chronic oedema), e.g. of the legs, is quite a common condition, which can cause a number of problems, including infections (cellulitis) in the swollen area and ulceration. It seems to be particularly common in people who are overweight but this has not been studied in detail. This study aims to address this gap in knowledge. It will take place in two stages, running in parallel to each other with different groups of patients. The first stage will determine how common persistent swelling is among patients attending weight management services at the Royal Derby Hospital and how it impacts on every day life. The second stage will determine whether weight loss surgery improves the swelling.

The results will inform future treatment guidelines for overweight patients who have swelling. They will also inform the design of future research that will investigate the effects of weight loss surgery in more detail, for example by testing out methods of measuring fluid changes in the legs.

All new patients attending the weight loss service will be eligible to take part in the first stage of the study, as long as they: give their informed consent to take part, and can speak English (or have someone with them who speaks English). Participants will not have had weight loss surgery previously. The Stage 1 assessment is expected to take about 40 minutes and consists of: a single clinical assessment for each participant to identify the presence of the swelling and its degree in each of the affected areas and, up to 3 questionnaires concerning their quality of life and mobility.

Patients attending the programme, who have been referred for bariatric surgery, will take part in the second stage of the study. Stage 2 will last approximately 13 months, during which time the participants will be assessed 4 times - once before surgery and at 3, 6, and 12-month intervals after surgery. Each Stage 2 assessment is expected to take about 50 minutes and consists of: a clinical assessment and up to 5 questionnaires.

DETAILED DESCRIPTION:
The clinical assessments included in both stages of the study will identify the presence and severity of swelling in each of the affected areas. Each assessment will consist of a clinical examination of the patient's legs and abdomen to look for swelling and changes in the skin associated with this.

Assessments carried out in Stage 1 will include bioimpedance and tissue dielectric constant (TDC) techniques.

* Bioimpedance measures the total fluid within a limb. This test passes an extremely small electrical current through the participant's body and measures the resistance to the flow of this current. The participant will not feel anything when the measurement is carried out as the current is very small, similar to the strength of a watch battery. If the participant is able to, the test will be undertaken with the participant lying down on an examination couch or sitting in a chair. Small stickers will be placed on the participant's hands and feet, and clips attached to these.
* The TDC measures fluid levels at different points. In order to record these fluid levels, a probe will be placed against the participants' skin on their feet, lower legs, and thighs.

Assessments carried out in Stage 2 will include bioimpedance, TDC, and also perometry (or measuring using a tape measure).

- This test measures the size and shape of the participants' legs, and can be undertaken by one of two methods depending on their mobility. If they need to stay in a chair or examination couch during the assessment, the size of their legs will be measured at different points using a tape measure. However, if possible, a device called a perometer will be used. Participants will be asked to stand with one leg in the frame of the perometer while it is moved up and down the leg. The frame contains lights which are used to measure the size and shape of the limb.

None of the assessments included in either stage should cause any pain or discomfort.

The questionnaires, which will be completed in both stages, concern the participants' quality of life and mobility.

* The EQ-5D questionnaire compares quality of life over time well and can assess the health utility of the participants. The EQ-5D scores can be used to calculate quality-adjusted life years.
* The GAD-7 (Generalised Anxiety Disorder 7-item Scale) and PHQ-9 (Patient Health Questionnaire - 9) questionnaires will be used to assess the anxiety/depression of the participants. Stage 1 participants will have completed these before their study assessments so the study team will obtain these results from their clinical records. Stage 2 participants will complete the questionnaires as part of the study assessments.
* The SF-36 questionnaire will assess the mobility of the participants and give general health-related quality of life scores.
* The LYMQOL questionnaire, which will only be given to participants who have oedema, is a validated, condition-specific, quality of life instrument. It can be used both: to assess lymphoedema of the limbs and as an outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have capacity to give informed consent.
* Ability to understand the assessment questionnaires in English.

Stage 1 - all patients accepted for referral. There are no co-morbidities that would exclude people.

Stage 2 - patients that undergo bariatric surgery.

Exclusion Criteria:

- Patients under the lower age limit of 18.

Stage 2 - By-Band-Sleeve study participants who are taking part in the randomisation part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 1 will assess patients attending the Tier 3 weight management programme at the Royal Derby Hospital, who are accepted for referral and provide informed consent to take part in the study.
  Stage 2 will assess patients attending the Tier 4 programme who undergo bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Stage 1 - Prevalence of chronic oedema - using a clinical assessment | 6 months
  This will be achieved using: a clinical assessment to identify the presence or absence of chronic oedema.
Stage 1 - Impact of chronic oedema - using a clinical assessment | 6 months
  This will be achieved using a clinical assessment to identify the degree of swelling in the affected areas.
Stage 1 - Impact of chronic oedema - using questionnaires | 6 months
  This will be achieved using a range of quality of life questionnaires to identify the impact that the swelling has on the participants.
Stage 2 - Definition of post-surgery changes in chronic oedema - using clinical assessments | Over 1 year, 6 months
  This will be achieved by serial clinical assessment measures over a 12-month follow up after surgery.

SECONDARY OUTCOMES:
Stage 1 - Comparison of quality of life - using questionnaires | 6 months
  The quality of life of participants with and without chronic oedema will be compared, using the scores from the quality of life questionnaires.
Stage 1 - Defining chronic oedema - using bioimpedance data | 6 months
  The bioimpedance data (measures total fluid within the legs) will be used to determine if the technique can define chronic oedema in this setting.
Stage 1 - Defining chronic oedema - using tissue dielectric constant data | 6 months
  The tissue dielectric constant data (measures fluid levels at different points) will be used to determine if the technique can define chronic oedema in this setting.
Stage 1 - Presence/severity of oedema - using questionnaires | 6 months
  The questionnaires will be used to collect data about the presence/severity of swelling of the patients. These will be important as they will help to determine the impact of chronic oedema on everyday life.
Stage 2 - Measuring oedema changes - using bioimpedance data | Over 1 year, 6 months
  The bioimpedance technique will be used to measure changes in the oedema from the baseline (pre-operative) measurement. The use of this technique will be validated by comparing the results with clinical assessment and limb volume measurements.
Stage 2 - Measuring oedema changes - using tissue dielectric constant data | Over 1 year, 6 months
  The tissue dielectric constant technique will be used to measure changes in the oedema from the baseline (pre-operative) measurement. The use of this technique will be validated by comparing the results with clinical assessment and limb volume measurements.
Stage 2 - Comparison over a 12-month period - comparing clinical assessments | Over 1 year, 6 months
  The clinical assessments [presence/severity of swelling and wounds (if present)] of the patients from their preoperative to their 12-month post-operative appointment will be compared in order to determine the impact of weight loss on chronic oedema. The effect sizes of these changes will be used to inform future study design and sample size calculation.
Stage 2 - Comparison over a 12-month period - comparing questionnaires | Over 1 year, 6 months
  The quality of life scores of the patients from their preoperative to their 12-month post-operative appointment will be compared in order to determine the impact of weight loss on chronic oedema. The effect sizes of these changes will be used to inform future study design and sample size calculation.
Stage 2 - Future sample size calculation - using recruitment data | Over 1 year, 6 months
  Recruitment data (the percentage of eligible patients who consent to take part in the study, and the number withdrawing or not completing the study follow-up) will be used to inform sample size calculation for the future study.

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan L Keeley, PhD, FRCP, Principal Investigator — University of Nottingham, School of Medicine
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be sent out after the study has ended to participants who request them.

REFERENCES:
- [Derived] Newman A, Keeley V, Pinnington L, Green C, Riches K, Franks PJ, Idris I, Moffatt CJ. Prevalence and Impact of Chronic Edema in Bariatric Patients: A LIMPRINT Study. Lymphat Res Biol. 2021 Oct;19(5):431-441. doi: 10.1089/lrb.2021.0055. PMID 34672794